CLINICAL TRIAL: NCT06046001
Title: AirWaze - Easy and Advanced Tools for CBCT Guided Lung Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XCY607-130895
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AirWaze (Experimental): AirWaze - easy and advanced tools for CBCT guided lung interventions
  Interventions: Device: AirWaze

INTERVENTIONS:
Device: AirWaze — AirWaze - easy and advanced tools for CBCT guided lung interventions

SUMMARY:
The goal of this clinical trial is to assess the overall usability of the Philips

AirWaze investigational device in patients indicated for CBCT-guided navigation bronchoscopy procedure. The main questions it aims to answer are to assess the:

* overall usability of the device
* accuracy of the tool-in-lesion confirmation scan Participants will undergo bronchoscopy with the new navigation device and additional confirmation scans. Follow-up visit at 7days will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of informed consent.
* ASA physical status between 1 and 3.
* Subject is willing and able to give written informed consent for clinical investigation participation prior to the procedure.
* Subject has a pulmonary lesion with an indication for diagnostic evaluation following current clinical guidelines and/or as decided by multi-disciplinary team consultation.
* Suitable for CBCT-guided endobronchial nodule biopsy under general anaesthesia.
* Pre-procedural (PET-)CT scan is available prior to the CBCT-NB intervention.

Exclusion Criteria:

* Aged 17 or younger at the time of informed consent.
* ASA physical status is equal to and greater than 4.
* Not willing or not able to give informed consent.
* Does not indicate diagnostic evaluation with navigation bronchoscopy.
* Not suitable for CBCT-guided endobronchial nodule biopsy via navigation bronchoscopy under general anaesthesia.
* There is no recent pre-procedural (PET-)CT scan available.
* Known bleeding disorders.
* Contra-indication for temporary interruption of the use of anticoagulant therapy, such as acenocoumarol, warfarin, therapeutic dose of low molecular weight heparins, clopidogrel, or analogues, NOACs).
* Known allergy for lidocaine or other allergies interfering with the procedure.
* Uncontrolled pulmonary hypertension.
* Recent and/or uncontrolled cardiac disease.
* Compromised upper airway (e.g. concomitant head and neck cancer or central airway stenosis for any reason such that endobronchial access is considered unsafe).
* Potentially confounding drug or device trial during the clinical study. Co-enrollment in concurrent trials may be allowed provided pre-approval is obtained from the Philips Clinical Study Manager.
* All vulnerable subjects, such as immune-compromised subjects, subjects lacking the capacity to provide consent, patients in emergencies, pregnant or breastfeeding women, or any other subject who meets exclusion criteria, according to applicable national laws, if any.
* Woman of childbearing potential who is known to be pregnant on admission.
* Any condition that in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the subject in the study.
* Subject is Philips employee or their family members residing with this Philips employee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
System Usability Score (SUS) | Pre-procedure and immediately after the procedure
  System Usability Score (SUS) of AirWaze investigational device. An average SUS of greater than 70 will indicate a good usability design of the AirWaze Software solution. The SUS will be measured per operator every 4 procedures. The questionnaire consists of a 10-item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. Minimum total score is 0 and maximum, 100.
Accuracy of the tool-in-lesion confirmation scan assessed by questionnaire "CBCT-FS compared to CBCT". | Immediately after the procedure
  Accuracy of the tool-in-lesion confirmation scan compared to the conventional scan based on questionnaire about tool-in-lesion definitions and usefulness of the scans to guide to the lesion (questionnaire "CBCT-FS compared to CBCT"). Image based tool-in-lesion confirmation accuracy of 90% will indicate that the CBCT-FS is postulated to be sufficient for navigation bronchoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Erik van der Heijden, Principal Investigator — Radboudumc Nijmegen, Netherlands
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No